CLINICAL TRIAL: NCT03327532
Title: Acute Heart Failure - COngestion Repeated Evaluation (AHF-CORE). Evaluation répétée de la Congestion au Cours d'Une Hospitalisation Pour Insuffisance Cardiaque aigüe
Brief Title: Acute Heart Failure - COngestion Repeated Evaluation (AHF-CORE)
Acronym: AHF-CORE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Pr. Nicolas GIRERD, Professor, Central Hospital, Nancy, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2017-A01455-48
Record Dates: First submitted 2017-09-06; First posted 2017-10-31 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Acute Heart Failure
Keywords: Acute Heart Failure; Congestion; Ultrasound
MeSH Terms: interventions — Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients hospitalized for acute heart failure (Experimental): One arm study.
  Patients hospitalized for acute heart failure will undergo the following evaluations:
  * Clinical examination centered on congestion
  * Cardiopulmonary and peritoneal ultrasound
  * Blood sample retrieved for biological assessment and biobanking
  * Telephone interview
  Interventions: Procedure: Clinical examination centered on congestion; Procedure: Cardio-pulmonary and peritoneal ultrasound; Biological: Blood sample retrieved for biological assessment and biobanking; Other: Telephone interview; Biological: Urinary sample retrieved for biological assessment and biobanking; Procedure: jugular and renal ultrasound (optional)

INTERVENTIONS:
Procedure: Clinical examination centered on congestion — Clinical examination centered on congestion will be performed within 72 hours of admission and before discharge from hospital
Procedure: Cardio-pulmonary and peritoneal ultrasound — Cardio-pulmonary and peritoneal ultrasound will be performed within 72 hours of admission and before discharge from hospital
Biological: Blood sample retrieved for biological assessment and biobanking — Blood sample collection will be performed within 72 hours of admission and before discharge from hospital
Other: Telephone interview — Telephone interview will be performed 3, 12 and 24 months after discharge from hospital
Biological: Urinary sample retrieved for biological assessment and biobanking — Urinary sample collection will be performed within 72 hours of admission and before discharge from hospital
Procedure: jugular and renal ultrasound (optional) — optional jugular and renal ultrasound performed within 72hours of admission and before discharge from hospital

SUMMARY:
The AHF-CORE study is a prospective, non-randomized, multicenter regional study.

The main objective of the AHF-CORE study is to identify congestion markers (clinical, biological and ultrasound) at the beginning and at the end of hospitalization for acute heart failure that are more strongly associated with the risk of all cause death or rehospitalization for acute heart failure within 3 months of hospital discharge.

Secondary objectives are:

* Quantify the variations in congestion markers between the beginning and end of hospitalization for acute heart failure.
* Assess the correlation between changes in congestion markers between the beginning and end of hospitalization.
* Identify the congestion markers at the beginning of hospitalization that are most strongly associated with residual congestion at the end of hospitalization.
* Identify the added value of ultrasound and biological markers of congestion in addition to clinical variables for the prediction of all-cause death or hospitalization for acute heart failure at 3 months after hospital discharge.
* Identify the association of ultrasound and biologic congestion markers assessed at admission and final discharge with NYHA class at 3 months after hospital discharge

DETAILED DESCRIPTION:
Congestion (clinical, biological and ultrasound evaluation) will be quantified at inclusion within 72 hours of admission and before hospital discharge.

Follow-up at 3 months of hospital discharge will be performed through telephone interviews. Vital status and rehospitalization status will be collected.

Throughout the study, patients will continue to be treated according to usual routine care, regardless of their level of congestion. There will be no modification of treatment according to the congestion data acquired within the setting of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized for left-sided or global acute heart failure due to exacerbation of chronic heart failure within 72 hours of admission to hospital
* Patients over 18 years old
* Person affiliated to or beneficiary of a social security plan
* Person informed about study organization and having signed the informed consent

Exclusion Criteria:

* Comorbidity for which life expectancy is ≤ 3 months
* Diagnosis of heart failure made less than 3 months prior to inclusion
* Exacerbation of heart failure attributed to acute ischemic stroke (acute coronary syndrome with or without ST segment elevation)
* Dialyzed patient (peritoneal dialysis or hemodialysis) and patients with glomerular filtration rate <15 ml / min / m2 at baseline
* History of pulmonary lobectomy or pneumonectomy
* Severe pulmonary or pleural disease preventing the reliable acquisition of pulmonary ultrasound images: severe emphysema, chronic pleurisy, pulmonary fibrosis
* Suspected cardiac amylose or proven cardiac amylose
* Woman of childbearing age without effective contraception
* Persons referred in articles L.1121-5, L.1121-7, L.1121-8 and L.1122-2 of the French Public Health Code: Pregnant, parturient or breastfeeding woman ; Minor person (non-emancipated) ; Adult person under legal protection (any form of public guardianship) ; Adult person incapable of giving consent and not under legal protection.
* Persons deprived of liberty for judicial or administrative decision
* Persons subject to psychiatric care under articles L.3212-1 and L.3213-1 of the French Public Health Code

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-02-13 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Rate of all-cause death | at 3 months after hospital discharge
  composite endpoint: rate of all-cause death, hospitalization for acute heart failure or day-hospital IV diuretics injection for acute HF during 24 months following the day hospitalization (with outcome 2 and 3)
Rate of rehospitalization for acute heart failure | at 3 months after hospital discharge
  composite endpoint: rate of all-cause death, hospitalization for acute heart failure or day-hospital IV diuretics injection for acute HF during 24 months following the day hospitalization (with outcome 1 and 3)
Rate of day-hospital or at-home IV diuretics injection for acute HF | at 3 months after hospital discharge
  composite endpoint: rate of all-cause death, hospitalization for acute heart failure or day-hospital IV diuretics injection for acute HF during 24 months following the day hospitalization (with outcome 1 and 2)

SECONDARY OUTCOMES:
Clinical congestion markers as assessed with the Ambrosy Score | at admission and at final discharge (an average of 10 days after admission)
  Clinical congestion markers as assessed with the Ambrosy Score at admission and at final discharge
Clinical congestion markers as assessed with the ASCEND score | at admission and at final discharge (an average of 10 days after admission)
  Clinical congestion markers as assessed with the ASCEND score at admission and at final discharge
Natriuretic peptides | at admission and at final discharge (an average of 10 days after admission)
  Natriuretic peptides at admission and at final discharge
Estimated plasma volume | at admission and at final discharge (an average of 10 days after admission)
  Estimated plasma volume at admission and at final discharge
Ultrasound congestion markers | at admission and at final discharge (an average of 10 days after admission)
  B lines, pleural effusion, E/e', DTE, TRV, VCI, Jugular diameter, renal venous blood flow pattern, peritoneal effusion
Residual congestion | at final discharge (an average of 10 days after admission)
  as defined as an Ambrosy score 3 or more and/or B-lines score 30 or more and/or an IVC>21 and IVC collapse with sniff <50%
NYHA class | 3 months after hospital discharge
  NYHA class (1, 2, 3, 4)
Rate of day-hospital for Intravenous diuretics administration for acute HF | 3, 12 and 24 months after hospitalization
  To identify the markers of congestion (clinical, biological, and ultrasonographic), at the end of hospitalization for ICA most strongly associated with the risk of intravenous administration of diuretics in day-hospital for ICA at 3,12, and 24 months after hospital discharge.
Rate of all-cause death | 12 and 24 months after hospitalization
  composite endpoint: rate of all-cause death, hospitalization for acute heart failure or day-hospital IV diuretics injection for acute HF during 24 months following day hospitalization (with outcome 12 and 13)
Rate of hospitalization for acute heart failure | 12 and 24 months after hospitalization
  composite endpoint: rate of all-cause death, hospitalization for acute heart failure or day-hospital IV diuretics injection for acute HF during 24 months following day hospitalization (with outcome 11 and 13)
Rate of day-hospital or in-home IV diuretics injection for acute HF | 12 and 24 months after hospitalization
  composite endpoint: rate of all-cause death, hospitalization for acute heart failure or day-hospital IV diuretics injection for acute HF during 24 months following day hospitalization (with outcome 11 and 12)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas GIRERD, MD,PhD, Principal Investigator — Centre d'Investigation Clinique 1433 module Plurithématique de Nancy
Locations (2):
- France (2):
  - CHR Metz-Thionville - Hôpital de Mercy, Metz, Lorraine
  - CHRU Nancy Hôpitaux de Brabois, Vandœuvre-lès-Nancy, Lorraine

IPD SHARING:
Plan to Share IPD: No